CLINICAL TRIAL: NCT06681051
Title: Effectiveness and Safety of OSTENIL® TENDON in the Treatment of Pain and Restricted Mobility in Tendon Disorders
Status: Recruiting | Type: Observational
Sponsor: TRB Chemedica AG (Industry)
Responsible Party: Sponsor
Other Study IDs: OTIPPE-PMCF-DE-2021
Record Dates: First submitted 2024-11-07; First posted 2024-11-08 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Tendinopathy
Keywords: tendinopathy; hyaluronan; tendon; hyaluronic acid
MeSH Terms: conditions — Tendinopathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- OSTENIL® TENDON: 2 injections of sodium hayluronate 2 % (40 milligrams (mg) / 2.0 millilitres (ml)) in weekly interval.
  Interventions: Device: OSTENIL® TENDON

INTERVENTIONS:
Device: OSTENIL® TENDON — OSTENIL® TENDON is a CE-certified viscoelastic solution intended for peritendinous or intrasheath injection, containing 2 % sodium hyaluronate from fermentation.

SUMMARY:
PMCF study to further substantiate the effectiveness and safety of OSTENIL® TENDON in the overall as well as indication-specific treatment of pain and restricted mobility in four different tendon disorders (patella tendon, peroneal tendon, medial epicondylus humeri and iliotibial band) in a real-life clinical setting when used according to the instructions for use.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged between 18 and 99 years
* Diagnosis of symptomatic tendinopathy (patella tendon, peroneal tendon, medial epicondylus humeri or iliotibial band)
* Physician's recommendation to use OSTENIL® TENDON prior to recruitment
* Signed informed consent

Exclusion Criteria:

* Presence of any contra-indication or precautionary condition listed in the instructions for use, i.e.,

  * Ascertained hypersensitivity to any of the OSTENIL® TENDON constituents
  * Known pregnancy or breast feeding
  * Acute trauma
* Use of the following treatments (the given time intervals refer to the date of inclusion):

  * Local* OSTENIL® TENDON or other hyaluronic acid (HA) treatment within the last 6 months
  * Local* platelet-rich plasma (PRP) treatment within the last 3 months
  * Local* corticosteroid treatment (without time restriction)
  * Local* extracorporeal shock wave therapy (ESWT) within the last 4 weeks
  * Local* phytotherapy (e.g., Traumeel®) within the last 4 weeks
  * Local* surgical intervention (without time restriction)
  * Systemic corticosteroid treatment within the last 4 weeks
  * Repeated use of non-steroidal anti-inflammatory drugs (NSAID) and/or other analgesics within the last week
  * Physiotherapy (therapeutic exercises and physical therapy), ortheses, transcutaneous electrical nerve stimulation (TENS) or acupuncture within the last week
* Diagnosis of chronic inflammatory disease (e.g. rheumatoid arthritis, Bechterew disease, Crohn's disease, etc.) prior to inclusion
* Participation in a clinical investigation within the last 6 months
* Vulnerable patient (individual who is unable to fully understand all aspects of the study that are relevant to the decision to participate, or who could be manipulated or unduly influenced as a result of a compromised position, expectation of benefits or fear of retaliatory response [including persons needing legally designated representatives, illiterate persons or persons with insufficient knowledge of local language])

(* local refers to the treatment of the study-relevant tendon)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years of age with symptomatic tendinopathy (patella tendon, peroneal tendon, medial epicondylus humeri or iliotibial band) and a recommendation for OSTENIL® TENDON treatment.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change of pain intensity 3 months after end of treatment compared to baseline (visual analogue scale) | Baseline compared to week 12 after the end of treatment.
  Evaluation of pain intensity by the patient on a 100 mm visual analogue scale. 100 mm equals the worst pain.

SECONDARY OUTCOMES:
Change of Upper -/ Lower Extremity Functional Scale compared to baseline | Baseline compared to week 1 as well as weeks 4, 12 and 24 after the end of treatment.
  Indication specific patient questionnaire to assess effectiveness of treatment on a 5-point Likert scale (range: 0 = extreme difficulty to perform activity to 4 = no difficulty).
Change of pain intensity compared to baseline (visual analogue scale) | Baseline compared to week 1 as well as weeks 4 and 24 after the end of treatment.
  Evaluation of pain intensity by the patient on a 100 mm visual analogue scale. 100 mm equals the worst pain.
Change of patient-reported outcome measures (PROM) | Baseline (except satifaction with treatment), week 1 and weeks 4, 12 and 24 after the end of treatment.
  Patient questionnaire to assess the following aspects (100 mm visual analogue scale; 100 mm equals a worse outcome): pain, global and tendon-associated quality of life, daily activities, clinical global impression, mobility and satisfaction with treatment (note: not assessed at baseline)
Change of investigator-reported outcome measures | Baseline (except satisfaction with treatment), week 1 and weeks 4, 12 and 24 after the end of treatment.
  Investigator inquiry to record the perception of the physician of the following aspects (100 mm visual analogue scale; 100 mm equals a worse outcome):
  clinical global impression regarding the clinical severity of the tendinopathy and satisfaction with the treatment (note: not assessed at baseline)
Degree of tendinopathy | Baseline, week 1 and weeks 4, 12 and 24 after the end of treatment
  Evaluation of tendinopathy symptoms by the patient by rating tendon pain in the context of a patient-defined task that usually elicits pain (4 stages; 4 equals a worse outcome)
Incidence of Adverse Events with (possible/probable) causal relationship with the device or application procedure | Up to week 24 after the end of treatment.
Incidence of Serious Adverse Events with (possible/probable) causal relationship with the device or application procedure | Up to week 24 after the end of treatment.
Incidence of (Presumably) serious incidents | Up to week 24 after the end of treatment.
Incidence of Device Deficiencies | Up to week 24 after the end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Olaf Neubert, Dr. med., Principal Investigator — Orthopädie am Kiesteich
Locations (5):
- Germany (5):
  - Orthopädische Gemeinschaftspraxis ÜBAG, Berlin, State of Berlin
  - ATOS MVZ meviva Berlin, Berlin
  - Orthopädie am Kiesteich, Berlin
  - Orthopädie Dr. Bentzin, Berlin
  - Orthopädische Praxis Dr. Fischer, Potsdam

IPD SHARING:
Plan to Share IPD: No
Proprietary company data will not be shared externally.